CLINICAL TRIAL: NCT05954351
Title: PRactice of Ventilation and Adjunctive Therapies in COVID-19 Patients; What is the Optimal Ventilation Strategy in Critically Ill COVID-19 Patients, in Particular PEEP and the Moment of Switch to Pressure Support?
Brief Title: PRactice of Ventilation and Adjunctive Therapies in COVID-19 Patients.
Acronym: PRoVAcT-COVID
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Professor Dr. Marcus J. Schultz, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Other Study IDs: PRoVAcT-COVID
Record Dates: First submitted 2023-07-19; First posted 2023-07-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PRactice of Ventilation and Adjunctive Therapies in COVID-19 Patients. An observational study of ventilation practice and adjunctive therapies in critically ill, invasively ventilated COVID-19 patients during the first and second surge of COVID-19 in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* receiving invasive ventilation or high-flow nasal oxygen for COVID-19 for SARS-CoV-2
* admitted to one of the ICUs of the participating hospitals

Exclusion Criteria:

* none

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: invasively ventilation COVID-19 patients, admitted between March 1 to June 1, 2020, and October 1 to December 31, 2020, to one of the 22 participating ICU's in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 2465 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
ICU mortality | 90 days from inclusion

SECONDARY OUTCOMES:
Duration of ventilation | 90 days from inclusion
28-day ventilator free days | 90 days from inclusion
28-day, 90-day mortality | 90 days from inclusion
ICU and hospital length of stay | 90 days from inclusion

OTHER OUTCOMES:
Acute kidney injury | 90 days from inclusion
duration of ventilation in survivors | 90 days from inclusion
use of muscle paralysis | 90 days from inclusion
vasopressor or inotrope administration | 90 days from inclusion
occurrence of tracheostomy | 90 days from inclusion
pneumothorax and thromboembolic complications | 90 days from inclusion
use of immunomodulating drugs | 90 days from inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided